CLINICAL TRIAL: NCT07381868
Title: Social Media Psychosocial Support Group to Reduce Alcohol Consumption in Women: a Pilot Randomized Controlled Trial
Brief Title: Social Media Psychosocial Support Group in Reducing Alcohol Consumption
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Women Alcohol Reduction
Record Dates: First submitted 2025-12-17; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-09

CONDITIONS: Alcohol; mHealth Intervention
Keywords: psychosocial support; alcohol consumption; adult women; social media; reduce alcohol intake
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conrtol group (Active Comparator): Participatns in the control group will receive alcohol brief intervention according to their AUDIT score at baseline and 4 weeks 1-to-1 health education messages.
  Interventions: Behavioral: Brief alcohol use counselling and health education
- Intervention group (Experimental): A 4-week psychological support group for interactive counselling will be provided to encourage reducing alcohol consumption. MHealth messages will also be provided according to the stages of change for alcohol use.
  Interventions: Behavioral: mHealth-based motivational counselling; Behavioral: Brief alcohol use counselling and health education; Behavioral: Social media group support with engagement management

INTERVENTIONS:
Behavioral: mHealth-based motivational counselling — The mHealth intervention will be delivered via the most popular instant messaging app in Hong Kong (WhatsApp). A total of 12 instant messages of six themes in multi-media formats, including text, pictures, animation, and short videos, will be sent to the participants according to the stages of change for alcohol use. Pre-contemplation: provide information about the risks of drinking; Contemplation: Emphasize the benefits of reduction and quitting, discuss alcohol problems and achievable goals for reduction or quitting; Preparation: discuss goal and give advice and encouragement; Action: review advice and provide encouragement; and Maintenance: give encouragement.Using a more personalized approach, the messages will be tailored to the participants' motivation, intention to quit and other quitting patterns collected at baseline. Real-time conversations could be initiated by participants themselves, triggered by regular messages, or through prompt inquires.
  Arms: Intervention group
Behavioral: Brief alcohol use counselling and health education — After randomization and baseline data collection, participants will be linked to an experienced behavior counsellor and to receive a brief alcohol use counselling with health education, including health risks in alcohol use, advice to reduce alcohol consumption and available alcohol use services in Hong Kong with self-help psychoeducational materials. Guided by WHO, personal feedback will be provided according to Alcohol Use Disorders Identification Test (AUDIT) score: 8-15 indicates at-risk for alcohol use, 16-19 indicates potentially harmful or hazardous drinking, and ≥20 indicates alcohol dependence. For subjects with potential risky drinking (3-8), AUDIT score will be explained and readiness to change drinking habits will be assessed.
Behavioral: Social media group support with engagement management — The behavior counsellor will invite the participants to join a psychological support group for interactive counselling. Counsellor will lead the discussion and provide counselling according to the stages of change for alcohol use. Pre-contemplation: provide information about the risks of drinking; Contemplation: Emphasize the benefits of reduction and quitting, discuss alcohol problems and achievable goals for reduction or quitting; Preparation: discuss goal and give advice and encouragement; Action: review advice and provide encouragement; and Maintenance: give encouragement. Participants will be encouraged to interact with counsellor on any concerns about healthy lifestyle, mood fluctuation, and other ways to deal with cravings.
  Arms: Intervention group

SUMMARY:
This proposed study aims to develop and examine the feasibility, acceptability, and preliminary effectiveness of a proactive intervention model that combines brief psychological counselling, Ecological Momentary Assessment (EMA) and social media psychosocial support group to reduce alcohol consumption in women.

DETAILED DESCRIPTION:
Targeted participants are adult women with a total a total score≥3 in Alcohol Use Disorders Identification Test - Consumption (AUDIT-C). Sixty participants will be actively recruited from the social media platform in Hong Kong.

This study will be a two-arm (allocation ratio:1:1; permutated block size of 2, 4, and 8), single blinded, parallel, pilot randomized controlled trial (RCT) with follow-ups at 4, 8, and 12 weeks post-enrollment using consolidated standards of reporting (CONSORT) to evaluate the effectiveness of the intervention. The control group will receive an evidence-based intervention composed of brief psychological counselling and health education, 4-week EMA and social media psychosocial support group, guided by comprehensive assessment. Surveys will be collected via telephone. Semi-structured individual telephone or face-to-face indepth interviews will be conducted with the participants in the intervention group to understand the experience and the perceptions towards the EMA data collection and ocial media psychosocial support group intervention on alcohol consumption.

The clinical outcome of this study will be the difference in the alcohol consumption, anxiety and depressive levels, stress levels, and family well-being between the two groups at 4, 8, and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (age 18+),
* Had a total score ≥3 in AUDIT-C [suggesting at-risk drinkers (i.e., binge drinking)]( potential distress symptoms),
* Able to read and understand Chinese and use an instant messaging app weekly

Exclusion Criteria:

* Women who are undergoing psychiatric/psychological treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Alcohol use | 4-, 8-, and 12-weeks after enrollment
  Alcohol use is measured by the Alcohol Use Disorders Identification Test (AUDIT) scale. It is a standardized, 10-item self-report screening instrument developed by the World Health Organization (WHO) to identify hazardous alcohol consumption, harmful drinking behaviors, and alcohol use disorders (AUDs). Respondents rate each item on a 5-point Likert scale (0 = never to 4 = daily or almost daily), with total scores ranging from 0 to 40. The higher the score, the greater the risk of individual alcohol abuse and dependence. Established cutoff values guide interpretation: Scores 0-7: Generally indicates low-risk or abstinence. Scores 8-14: Suggests hazardous or harmful alcohol use. Scores 15-19: Indicates a high level of harmful alcohol use. Simple advice and periodic review are advised. Scores 20-40: Suggests a likely alcohol dependence syndrome and the need for further diagnostic evaluation and specialist treatment consideration.

SECONDARY OUTCOMES:
Anxiety | 4-, 8-, and 12-weeks after enrollment
  The Generalized Anxiety Disorder Scale (GAD-7) is a 7-item self-reporting scale that evaluates the frequency and severity of anxious thoughts and behaviors during the last 2 weeks. Items are based on the diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) criteria and scored from 0 (not at all) to 3 (nearly every day). Total scores range from 0 to 21, with established cutoff values for interpreting severity: 0-4 (minimal anxiety), 5-9 (mild anxiety), 10-14 (moderate anxiety), and 15-21 (severe anxiety).
Depressive symptoms | 4-, 8-, and 12-weeks after enrollment
  The Patient Health Questionnaire-9 (PHQ-9) is a self-reporting questionnaire comprising 9 items that evaluate the frequency and severity of depressive symptoms during the last 2 weeks (e.g., "Little interest or pleasure in doing things", "Feeling down, depressed, or hopeless"). Responses are scored on a 4-point Likert scale (0 = not at all to 3 = nearly every day), with total scores ranging from 0 to 27. Scores are typically interpreted as follows: 0-4 (minimal symptoms), 5-9 (mild depression), 10-14 (moderate depression), 15-19 (moderately severe depression), and 20-27 (severe depression).
Stress | 4-, 8-, and 12-weeks after enrollment
  This project measured the participants' stress level by using the Perceived Stress Scale (PSS-10). This is a ten-item scale that measures how often stressful events occurred the last month using a 5-point Likert scale from 'Never' to 'Very Often'(0 = never to 4 = very often). Total scores range from 0 to 40, where higher scores indicate higher levels of perceived stress. An example of an item was: "How often have you been able to control irritations in your life?"
Perceived family well-being | 4-, 8-, and 12-weeks after enrollment
  Perceived family well-being will be measured by the Family Apgar Scale. The scale comprises 5 core items that measure key dimensions of family well-being: adaptability (ability to cope with crises), partnership (shared decision-making and mutual support), growth (encouragement of individual development), affection (expression of warmth and care), and resolve (ability to solve conflicts effectively). Respondents rate each item on a 3-point Likert scale (0 = hardly ever to 2 = almost always), yielding a total score ranging from 0 to 10. Scores are interpreted as follows: 7-10 indicates healthy family functioning, 4-6 suggests moderate family dysfunction, and 0-3 signifies severe family dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Public Health, The University of Hong Kong, 18/F, Metro South Tower 1, 39 Wong Chuk Hang Road, Wong Chuk Hang, 999077, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No